CLINICAL TRIAL: NCT01410825
Title: Pilot and Feasibility Study of Hematopoietic Stem Cell Gene Transfer for the Wiskott-Aldrich Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Williams (Other)
Responsible Party: Sponsor-Investigator, David Williams, Chief of the Division of Hematology/Oncology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHB-P00000148
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: WAS; Wiskott; Gene Transfer; Gene Therapy
MeSH Terms: conditions — Wiskott-Aldrich Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gene transfer (Experimental): Open label single arm study
  Interventions: Biological: Retrovirus-mediated gene transfer

INTERVENTIONS:
Biological: Retrovirus-mediated gene transfer — Two procedures: 1) Bone marrow harvest from the patient's posterior iliac crests or collection of peripheral blood stem cells via apheresis procedure. 2) One time infusion of patient's transduced bone marrow cells.

SUMMARY:
The Wiskott-Aldrich Syndrome (WAS) is an inherited disorder that results in defects of the blood and bone marrow. It affects boys because the genetic mistake is carried on the X chromosome. Normal people have blood cells called platelets that stop bleeding when blood vessels are damaged. Boys with WAS have low numbers of platelets that do not function correctly. Boys with WAS are thus at risk for severe life-threatening bleeding. A normal immune system is made of special blood cells called white blood cells, which protect against infection and also fight certain types of cancer. In WAS, these white blood cells don't work as well as they should, making these boys very susceptible to infections and to a form of blood cancer known as lymphoma. The abnormal white blood cells of patients with WAS also cause diseases such as eczema and arthritis. Although WAS can be mild, severe forms need treatment as early as possible to prevent life-threatening complications due to bleeding, infection and blood cancer.

Over the past decade, investigators have developed new treatments based on the investigators knowledge of the defective gene causing WAS. The investigators can now use genes as a type of medicine that will correct the problem in the patient's own bone marrow. The investigators call this process gene transfer. The procedure is very similar to a normal bone marrow transplant, in that the old marrow is killed off using chemotherapy, but is different because the patient's own bone marrow is given back after it is treated by gene transfer. This approach can be used even if the patient does not have any matched donors available and will avoid problems such as GVHD and rejection. The investigators wish to test whether this approach is safe and whether gene transfer will lead to the development of a healthy immune and blood system.

DETAILED DESCRIPTION:
Wiskott-Aldrich syndrome (WAS) (OMIM 301000) is a rare X-linked immunodeficiency caused by mutations in a single gene, WAS, mapping to Xp11.22-Xp11.3 and coding for the Wiskott-Aldrich Syndrome Protein (WASP) 1. WASP is a critical regulator of actin signaling with expression limited to hematopoietic cells, and thus is required for multiple functions including T cell activation, dendritic cell migration and podosome formation, and B cell terminal development and function. WAS is characterized by microthrombocytopenia, recurrent infections, eczema and associated with a high incidence of auto-immunity and of lymphoid malignancies. Classic or severe WAS, is generally observed in patients with nonsense mutations or insertions/deletions resulting in frameshift or splice-site mutations or missense mutations and resulting in unstable protein 2. With few exceptions, WASP-negative patients have classical disease. Affected patients have a severely reduced life expectancy.

Currently, the only curative option for WAS patients is hematopoietic stem cell transplantation (HSCT). This treatment is most successful when an HLA-identical sibling or matched unrelated donor is available and results in correction of microthrombocytopenia and immune dysfunction, even when stable mixed chimerism occurs. However, even patients undergoing matched HSCT can suffer from considerable morbidity and mortality due to graft versus host disease (GVHD) and many patients lack an HLA-identical donor. The outcome of mismatched related HSCT is consistently poor with survival of approximately 50%. Gene transfer is an attractive alternative treatment for WAS. Successful gene transfer using autologous gene-corrected HSC would overcome clinical complications linked to GVHD and its treatment. Furthermore, in contrast to allogeneic HSCT, gene transfer would not be limited by the availability of compatible donors. Several lines of evidence indicate that partial reconstitution with gene corrected cells may be sufficient to ameliorate the disease.

We propose here a Pilot and Feasibility study of ex vivo gene transfer using a lentiviral vector (LV) to transduce autologous bone marrow derived CD34+ HSC. Cells will be infused into patients conditioned with cytoreductive chemotherapy. Our collaborating investigators in Europe have developed a LV encoding the human WAS cDNA under control of the WAS promoter and pseudotyped with the Vesicular Stomatitis Virus glycoprotein (VSVg) envelope. This w1.6_hWASP_WPRE (VSVg) LV (abbreviated as w1.6W) has been shown to be efficacious in both in vitro and in vivo preclinical models. Safety including cellular toxicity, insertional mutagenesis and tumor formation has been studied by a number of methods including: 1) a sensitive in vitro transformation assay, 2) toxicity studies in transduced human CD34+ cells, 3) examination of the insertional pattern in transduced murine cells, and 4) long-term observation and secondary transplant studies in mice. In the United States, we plan to enroll 5 boys with classic WAS who lack a matched related or unrelated donor. Parallel studies (not under our Investigational New Drug application) using the same LV produced in the same facility, Genethon, will be conducted in London, UK (5 subjects) and Paris, France (5 subjects). The primary objective will be to demonstrate feasibility and safety. The secondary objective will be to assess therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed molecular diagnosis by DNA sequencing and either

   1. absence of the WAS protein by flow cytometry OR
   2. clinical score 3-5
2. Age 3 months to 35 years
3. For subjects < 5 years of age:

   1. Lack of HLA-genotypically identical bone marrow donor.
   2. Lack of a 9/10 or 10/10 molecularly HLA-matched unrelated donor after 3 months of searching.
   3. Lack of a 6/6 molecularly HLA-matched cord blood donor of adequate cell number after 3 months of searching
4. For subjects 5 years of age or older:

   a.Lack of HLA-genotypically identical bone marrow donor.
5. Subjects who have undergone allogeneic transplant previously must additionally have:

   1. Failure defined as <5% donor T cell engraftment and
   2. Contraindication to re-use of the same donor due to severe GVHD or non-availability.
6. Parental/guardian/patient signed informed consent
7. Willingness to return for follow-up during the 5 year study period.
8. Adequate organ function and performance status

   1. Performance status ≥50% (Lansky play for age <16 years, Karnofsky for age ≥16 years)
   2. Left ventricular ejection fraction >40% or shortening fraction >25%
   3. Bilirubin ≤ 2.0 mg/dL
   4. Measured creatinine clearance or GFR by nuclear medicine study ≥40 ml/min/1.73 m2
   5. DLCO (corrected for hemoglobin), FEV1, FVC >50% of predicted; if age < 7 years, then oxygen saturation >92% on room air

Exclusion Criteria:

1. Contraindication to bone marrow harvest, or to administration of conditioning medication.
2. Known positive HIV serology or HIV nucleic acid testing.
3. Other uncontrolled infection.
4. Active malignancy other than EBV lymphoproliferative disease.
5. Known myelodysplasia of the bone marrow or abnormal bone marrow cytogenetics
6. Congenital cardiac disease with congestive heart failure
7. Oxygen dependence at baseline
8. Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful study completion. This may include but is not limited to:

   * Severe deterioration of clinical condition after collection of cells but before infusion of transduced cells
   * Documented refusal or inability of the family to return for scheduled visits
   * Other concerns about unwillingness or inability to comply with protocol requirements
   * Unforeseen rare circumstances such as sudden loss of legal guardianship

Ages: 3 Months to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Safety of infusion of transduced cells | 5 Years
  Safety of infusion of transduced cells as rescue of hematopoiesis after conditioning (hematopoietic recovery as assessed by absolute neutrophil count (ANC) above 0.5 x 109 /l for three consecutive days, achieved within 6 weeks following infusion).
Engraftment of genetically corrected T cells | 5 Years
  Engraftment of genetically corrected T cells in peripheral blood (as assessed by evidence of vector sequences in >1% of CD3+ T cells) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whangbo, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labrosse R, Chu JI, Armant MA, Everett JK, Pellin D, Kareddy N, Frelinger AL, Henderson LA, O'Connell AE, Biswas A, Coenen-van der Spek J, Miggelbrink A, Fiorini C, Adhikari H, Berry CC, Cantu VA, Fong J, Jaroslavsky J, Karadeniz DF, Li QZ, Reddy S, Roche AM, Zhu C, Whangbo JS, Dansereau C, Mackinnon B, Morris E, Koo SM, London WB, Baris S, Ozen A, Karakoc-Aydiner E, Despotovic JM, Forbes Satter LR, Saitoh A, Aizawa Y, King A, Nguyen MAT, Vu VDU, Snapper SB, Galy A, Notarangelo LD, Bushman FD, Williams DA, Pai SY. Outcomes of hematopoietic stem cell gene therapy for Wiskott-Aldrich syndrome. Blood. 2023 Oct 12;142(15):1281-1296. doi: 10.1182/blood.2022019117. PMID 37478401